CLINICAL TRIAL: NCT02694848
Title: Clinical Study of Combination Therapy for Angina of Coronary Heart Disease With Aspirin and Salvianolate Injection Based on Population Pharmacokinetics and Therapeutic Effect:A Randomized, Controlled Trial
Brief Title: Clinical Study of Combination Therapy for Angina of Coronary Heart Disease With Aspirin and Salvianolate Injection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other); Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other); General Hospital of Beijing PLA Military Region (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xie Yanming, Director of institute of traditional Chinese medicine (TCM) clinical and basic medical science, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EBM
Record Dates: First submitted 2016-02-14; First posted 2016-03-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Angina
MeSH Terms: conditions — Angina Pectoris | interventions — salvianolate; Aspirin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Salvianolate injection group (Other): Salvianolate injection,intravenously infusion,0.2g/time,once a day;other routine treatment according to the condition of the disease
  Interventions: Drug: Salvianolate injection
- Aspirin group (Active Comparator): Aspirin,oral administration method,0.1g/time,once a day;other routine treatment according to the condition of the disease
  Interventions: Drug: Aspirin
- Salvianolate injection and aspirin group (Experimental): Salvianolate injection,intravenously infusion,0.2g/time,once a day;aspirin,oral administration method,0.1g/time,once a day;other routine treatment according to the condition of the disease
  Interventions: Drug: Salvianolate injection; Drug: Aspirin

INTERVENTIONS:
Drug: Salvianolate injection — Traditional Chinese medicine injection，a kind of innovative drugs developed by Shanghai institute of materia medica, Chinese academy of sciences after 13 years of research and development.the content of magnesium acetate was 80%, and the other 20% were magnesium acetate.It has the function of promoting blood circulation,removing blood stasis and blood stasis,and is used for treating coronary heart disease with stable angina pectoris.
  Arms: Salvianolate injection and aspirin group; Salvianolate injection group
Drug: Aspirin — Molecular chemical formula: C9H8O4,molecular structure type: CH3COOC6H4COOH. It has the role of anti thrombosis In vivo, and it can inhibit the release of the platelet reaction, inhibit platelet aggregation, which is related to the reduction of TXA2 generation. Clinically itused to prevent the onset of cardiovascular and cerebrovascular diseases.
  Arms: Aspirin group; Salvianolate injection and aspirin group

SUMMARY:
To evaluate the therapeutic evaluation of combination therapy with aspirin and salvianolate injection based on the population pharmacokinetics and TEG.A prospective, multicenter, randomized, controlled clinical trial is used.A total of 120 patients will be recruited and will be divided into three groups,respectively salvianolate injection group,aspirin group and salvianolate injection and aspirin group，and the course of treatment is 10 days.

DETAILED DESCRIPTION:
1. Effectiveness evaluation:Primary Outcome Measure:Change of TEG（R time, K time, α angle, MA,CI,TPI）.Secondary Outcome Measures: Change of symptom score of the Seattle Angina Questionnaiire(SAQ).Change of ECG abnormalities.Change of score of traditional Chinese medicine(TCM) symptom curative effect rating scale. Change of platelet aggregation measured by light transmittance aggregometry(LTA).Change of serum lipids（TC、TG、HDL-C、LDL-C）.Change of fasting blood glucose.Population pharmacokinetics test(the detection of the blood concentration of magnesium lithospermate B and salicylic acid).
2. Safety evaluation:Change of PT,APTT,TT,FIB.Adverse events.Change of basic life sign.Gastrointestinal symptoms.Change of stool routine.Change of routine blood test.Change of urine routine.Change of liver function.Change of renal function.Change of fecal occult blood.
3. Number of participants:120 participants will be divided into three groups, the salvianolate group (n=40), the aspirin group(n=40) and the combination therapy group of salvianolate injection and aspirin(n=40).
4. Interventions:salvianolate injection group: salvianolate injection, intravenously infusion,0.2g/time, once a day; other routine treatment according to the condition of the disease.Aspirin group: aspirin, oral administration method,0.1g/time, once a day; other routine treatment according to the condition of the disease.Salvianolate injection and aspirin group: salvianolate injection, intravenously infusion,0.2g/time, once a day; aspirin, oral administration method,0.1g/time, once a day; other routine treatment according to the condition of the disease.
5. Course of treatment：10 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 35-75 years old
* Grade II diagnostic criteria for chronic stable angina pectoris
* Diagnostic criteria of blood stasis type
* Signed informed consent

Exclusion Criteria:

* Drug allergy to the test
* There is a family or personal history of hemorrhagic disease
* Platelet count < 100 * nine times square 10/L or > 450 *nine times square 10/L
* Hemoglobin < 90g/L
* ALT, AST higher than the upper limit of 2 times, BUN, Cr higher than the upper limit
* Drugs such as the use of clopidogrel, clopidogrel, Hua Falin or heparin in the last 2 weeks to take blood circulation drugs or other antiplatelet, anticoagulant or non steroidal anti-inflammatory drugs
* Heart failure three degrees, two degrees in patients with heart failure
* A history of trauma or surgery in the past 2 weeks
* Combined coronary heart disease myocardial infarction and cerebral blood vessels, liver, kidney, hematopoietic system severe primary disease, malignant tumor, mental disease patients, as well as hyperthyroidism, cervical spondylosis, stomach and esophageal reflux and other patients with chest pain
* Organ transplantation, AIDS, long-term use of immunosuppressive agents and other immune deficiency
* Pregnant or lactating women
* Other clinical trial participants who are taking part in the evaluation of the results of this study

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change of thromboela-stogram（R time,K time,α angle,MA、CI、TPI） | Change from base line on the tenth day
  Thromboela-stogram(TEG) Is a reflection of the dynamic changes in blood coagulation (including the formation rate of fibrin, the dissolution of the state and the consistency of the solid, elastic degree) of the index: R time is the latency of the first fibrin plaque formation. K time is to assess the rate at which blood clots reach a certain level. The alpha angle is similar to the K time, but is more comprehensive than the K time, and is not affected by the low coagulation state. MA reflects the maximum amplitude of blood clots. CI is an integrated coagulation index.TPI is the index of platelet kinetics

SECONDARY OUTCOMES:
Change of symptom score of the Seattle Angina Questionnaiire(SAQ) | Change from base line on the tenth day
  SAQ includes 5 dimensions: the degree of physical activity limitation, the stable state of angina pectoris, the frequency of angina attack, the degree of treatment satisfaction, and the recognition of the disease
Change of ECG abnormalities | Change from base line on the tenth day
  ECG is the most common method of detection of myocardial ischemia and the diagnosis of angina pectoris
Change of score of Traditional Chinese Medicine(TCM) symptom curative effect rating scale | Change from base line on the tenth day
  It includes the description of scores of symptoms, signs of tongue and pulse related to blood stasis syndrome of diagnosis of traditional Chinese medicine
Change of platelet aggregation measured by light transmittance aggregometry(LTA) | Change from base line on the tenth day
  The method is widely recognized, and is even considered a gold standard
Change of serum lipids（TC、TG、HDL-C、LDL-C） | Change from base line on the tenth day
  Hyperlipidemia is one of the causes of angina. The measurement units of four indicators（TC、TG、HDL-C、LDL-C）are "mmol/L"
Change of fasting blood glucose | Change from base line on the tenth day
  It is one of the causes of angina(especially for patients with diabetes).The measurement unit is "mmol/L"
The blood concentration of magnesium lithospermate B | At the discretional two time points from the time point after treatment(0h,0.25h(15min),0.5h,0.75h(45min),1h,1.17h(70min),1.33h(80min),1.67h(100min),2h,2.5h,3h,4h,5h,7h,9h,13h,25h)
  Population pharmacokinetics test is in order to study the relationship between the population pharmacokinetics and clinical outcome. Magnesium lithospermate B is the main effective components of Salvianolate injection.The detection of the blood concentration of magnesium lithospermate B from both salvianolate injection group and salvianolate injection and aspirin group is necessary.
The blood concentration of salicylic acid | At the discretional two time points from the time point after treatment(0h,0.5h,1h,1.5h,2h,2.5h,3h,4h,5h,6h,8h,9h,10h,12h)
  Population pharmacokinetics test is in order to study the relationship between the population pharmacokinetics and clinical outcome. Salicylic acid is a kind of metabolite of aspirin. The detection of the blood concentration of salicylic acid from both aspirin group and salvianolate injection and aspirin group is necessary.

OTHER OUTCOMES:
Change of PT | Change from base line on the tenth day
  An index to reflect the status of the extrinsic coagulation system
Adverse events | Change from base line on the tenth day
Change of basic life sign | Change from base line on the tenth day
  In the medical care system, body temperature, blood pressure and pulse are the most important and basic three physiological parameters of the vital signs
Gastrointestinal symptoms | Change from base line on the tenth day
Change of stool routine | Change from base line on the tenth day
  The stool routine includes stool properties, lipid droplets, and white blood cell count
Change of routine blood test | Change from base line on the tenth day
  The routine blood test includes white blood cell count, neutral cell ratio, lymphocyte ratio, single nuclear cell ratio, red blood cell count, hemoglobin, platelet count
Change of urine routine | Change from base line on the tenth day
  The urine routine includes white blood cell count, red blood cell count,urine protein,urine sugar
Change of liver function | Change from base line on the tenth day
  The liver function includes glutamic-pyruvic transaminase,glutamic-oxalacetic transaminase
Change of renal function | Change from base line on the tenth day
  The renal function includes creatinine,usea nitrogen
Change of fecal occult blood | Change from base line on the tenth day
  In order to monitor the safety of the digestive tract (if there is bleeding)
Change of APTT | Change from base line on the tenth day
  An index to reflect the status of endogenous coagulation system
Change of TT | Change from base line on the tenth day
  An index to reflect the time consuming from the fibrinogen into fibrin
Change of FIB | Change from base line on the tenth day
  An index to reflect the content of fibrinogen

CONTACTS AND LOCATIONS:
Overall Officials: Yanming Xie, Study Chair, Study Chair — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences
Locations (1):
- Xiyuan Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lyu J, Xue M, Li J, Lyu W, Wen Z, Yao P, Li J, Zhang Y, Gong Y, Xie Y, Chen K, Wang L, Chai Y. Clinical effectiveness and safety of salvia miltiorrhiza depside salt combined with aspirin in patients with stable angina pectoris: A multicenter, pragmatic, randomized controlled trial. Phytomedicine. 2021 Jan;81:153419. doi: 10.1016/j.phymed.2020.153419. Epub 2020 Dec 10. PMID 33360345